CLINICAL TRIAL: NCT00501163
Title: Direct Measurements of Cardiometabolic Risk in Treated Schizophrenia Patients
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0574
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia; Cardiovascular Disease
Keywords: Schizophrenia; Cardiovascular; Risk
MeSH Terms: conditions — Schizophrenia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Participants will be asked to do the following:

1. A screening session in which you will take part in a diagnostic interview that will take about 2-3 hours to complete and will address your medical history. If you've recently participated in one of Dr. Haupt's or Dr. Newcomer's studies (HRPO #03-1281, 01-0134, or 04-0191) you may not have to complete this screening interview.
2. An ultrasound test of your heart and blood vessels where an ultrasound machine will use sound waves to create images that allow the main blood vessels in your neck to be examined. You will be lying down for the procedure, and a colorless gel will be applied to the side of your neck where the handheld probe (called a transducer) will be placed. The transducer will then be gently moved over each side of your neck. This procedure will take approximately 30 minutes.
3. A magnetic resonance image (MRI) study where the amount of fat in your liver will be measured. The MRI involves having your body painlessly scanned inside a tubular machine, while lying on a table for about 45 minutes.
4. Some routine blood tests to assess glucose (sugar) and lipid (fat) control and liver function, as well as an additional hepatitis screen if you have a history of hepatitis. You will go to the Intensive Research Unit (IRU) or Clinical Trials Unit (CTU) after an 8 to 10-hour overnight fast (except water). Approximately 42 ml (3 tablespoons) of blood will be obtained from you, and you will also have your height, weight, blood pressure, and waist and hip measurements taken. This will take approximately one hour.
5. A dual energy x-ray absorptiometry (DEXA) scan to measure your body fat and body muscle content. The DEXA scan involves lying on a table in a private room wearing a hospital gown for about 15 minutes while a machine silently measures the amount of fat in your body. The DEXA scan is part of the research study and gives the researcher a picture of how much fat is in your body.

DETAILED DESCRIPTION:
In comparison to the general population, major mental illness is associated with higher rates of heart disease, stroke, and diabetes. These problems can result in a life span that can be up to 25 years shorter than in people without a major mental illness. This study uses established medical tests that can predict how you might be affected. The purpose of this study is to compare the risk for these disorders in people with schizophrenia with the risk for these disorders in other people without schizophrenia.

ELIGIBILITY:
The inclusion criteria for the schizophrenia/schizoaffective group are: i) aged 18-55 years; ii) otherwise healthy and meets DSM-IV criteria for schizophrenia, any type, or schizoaffective disorder iii) able to give informed consent.

The inclusion criteria for children are: i) age 10-18 years; ii) otherwise healthy and meets DSM-IV criteria for one or more childhood-onset psychiatric disorder iii) able to give assent and have a guardian able to provide informed consent.

The inclusion criteria for the healthy controls are: aged 18-55 years; ii) otherwise healthy and do not meet DSM-IV criteria for any Axis I psychiatric illness; iii) able to give informed consent.

The exclusion criteria are: i) Any lifetime DSM-IV diagnoses of intravenous drug use or alcohol dependence, or if criteria for alcohol abuse were ever met, subject must have not met criteria for abuse within the last 12 months; ii) any history of hepatitis; iii) medications that can cause significant changes in hepatic function, glucose, or lipid metabolism, as determined by the investigator; iv) lipid lowering or glucose lowering medications; v) involuntary legal status (as per Missouri law); vi) pregnancy.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The inclusion criteria for the schizophrenia/schizoaffective group are: i) aged 18-55 years; ii) otherwise healthy and meets DSM-IV criteria for schizophrenia, any type, or schizoaffective disorder iii) able to give informed consent.
  The inclusion criteria for children are: i) age 10-18 years; ii) otherwise healthy and meets DSM-IV criteria for one or more childhood-onset psychiatric disorder iii) able to give assent and have a guardian able to provide informed consent.
  The inclusion criteria for the healthy controls are: aged 18-55 years; ii) otherwise healthy and do not meet DSM-IV criteria for any Axis I psychiatric illness; iii) able to give informed consent.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Haupt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States